CLINICAL TRIAL: NCT05883202
Title: Effect of the Abutment-Prosthesis Connection on Marginal Bone Loss and Gingival Sealing Around Dental Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Miguel Padial-Molina, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2622CEIH2022
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect® (Experimental): Restoration of multiple implants with a Connect® abutment between the implant and the prosthesis.
  Interventions: Device: Connect®
- Multi-unit (Active Comparator): Restoration of multiple implants with a conventional multi-unit abutment between the implant and the prosthesis.
  Interventions: Device: Multi-unit

INTERVENTIONS:
Device: Connect® — Restoration of multiple implants with a Connect® abutment between the implant and the prosthesis.
  Arms: Connect®
Device: Multi-unit — Restoration of multiple implants with a conventional multi-unit abutment between the implant and the prosthesis.
  Arms: Multi-unit

SUMMARY:
In dental implant restoration, available literature demonstrates the advantage of using tall abutments, with a change of diameter with respect to the implant and a conical internal connection in the abutment-implant gap. However, for multiple restorations, the abutment-prosthesis connection has not been studied in detail. The "multi-unit" systems, both standard and brand specific, have either a flat or butt joint or an cone. In any case, both are external connection systems. Recently, an internal-type abutment-prosthesis connection system has been developed. Although it is proving its usefulness in single restorations, its use in multiple restorations compared to traditional systems has not been studied.

Therefore, taking into account all of the above, the present study has the overall objective of analyzing marginal bone loss (MBL) and adaptation of soft tissues by comparing a multiple prosthesis system of the "external, flat" type versus an external system of the "internal, conical" type.

ELIGIBILITY:
Inclusion criteria:

* Kennedy class I or II (unilateral or bilateral free end) or III (posterior intermediate edentulous section) mandibular requiring 2 implants to restore at least 2 molars, 2 molars and 1 premolar, or 2 premolars and 1 molar.
* Possibility of placing a transgingival abutment at least 2 mm high.

Exclusion criteria:

* Need for simultaneous bone augmentation.
* Heavy smokers (>10 cigarettes/day).
* Uncontrolled type 1 or 2 diabetes (HgA1c>8).
* Known autoimmune or inflammatory disease.
* Serious blood disorders, such as hemophilia or leukemia.
* Local or systemic infection that may compromise normal healing (e.g., extensive periapical pathology).
* Liver or kidney dysfunction/failure.
* Currently receiving cancer treatment or within 18 months from completion of radio- or chemotherapy.
* Long-term history of oral bisphosphonates use (i.e., 10 years or more).
* History of intravenous bisphosphonates.
* Long-term (>3 months) history of antibiotics or drugs known to alter the inflammation and/or immunological system 3 months before inclusion.
* Severe osseous diseases (e.g., Paget disease of bone).
* Pregnant women or nursing mothers.
* Not able or not willing to follow instructions related to the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level | 1 year
  Peri-implant marginal bone level measured by standardized periapical radiography

SECONDARY OUTCOMES:
Peri-implant microbiome | 1 year
  Relative abundance of microbial species in the peri-implant sulcus evaluated by next-generation sequencing methods
Peri-implant inflammation | 1 year
  Concentration of pro-inflammatory markers in the peri-implant sulcus evaluated by multiplex techniques methods

OTHER OUTCOMES:
Soft-tissue volume | 1 year
  Three-dimensional volume of the soft tissue around the implants

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo-Moreno P, Leon-Cano A, Ortega-Oller I, Monje A, Suarez F, OValle F, Spinato S, Catena A. Prosthetic Abutment Height is a Key Factor in Peri-implant Marginal Bone Loss. J Dent Res. 2014 Jul;93(7 Suppl):80S-85S. doi: 10.1177/0022034513519800. Epub 2014 Mar 12. PMID 24621670
- [Background] Couso-Queiruga E, Tattan M, Ahmad U, Barwacz C, Gonzalez-Martin O, Avila-Ortiz G. Assessment of gingival thickness using digital file superimposition versus direct clinical measurements. Clin Oral Investig. 2021 Apr;25(4):2353-2361. doi: 10.1007/s00784-020-03558-0. Epub 2020 Aug 31. PMID 32865627